CLINICAL TRIAL: NCT04092725
Title: An Open-Label, Randomized, Two-Period, Crossover Study to Evaluate the Effect of Oral Doses of SCY-078 (Ibrexafungerp) on the Pharmacokinetics of Dabigatran Administered Orally to Healthy Subjects
Brief Title: Study to Evaluate the Effect of SCY-078 on the PK of Dabigatran in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scynexis, Inc. (Industry)
Collaborators: Clinical Network Services (CNS) Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SCY-078-108
Record Dates: First submitted 2019-09-03; First posted 2019-09-17 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Pharmacokinetics
Keywords: SCY-078; Dabigatran; Ibrexafungerp; Pharmacokinetics; Healthy Subjects
MeSH Terms: interventions — ibrexafungerp

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to a treatment sequence (AB or BA) in a crossover fashion with a minimum 10-day washout period between treatments.
  Treatment A = Single oral 150-mg dose of DAB on Day 1 AM. Treatment B = Twice daily (BID), every 12 hours (Q12H) oral doses of SCY-078 750 mg on Day 1 and Day 2; and single oral AM doses of SCY-078 750 mg on Day 3 and Day 4. On Day 3 a single 150-mg dose of DAB will be administered one hour after the AM dose of SCY-078.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Single oral 150-mg dose of DAB on Day 1 AM.
  Interventions: Drug: DAB
- Treatment B (Experimental): Twice daily (BID), every 12 hours (Q12H) oral doses of SCY-078 750 mg on Day 1 and Day 2; and single oral AM doses of SCY-078 750 mg on Day 3 and Day 4. On Day 3 a single 150-mg dose of DAB will be administered one hour after the AM dose of SCY-078.
  Interventions: Drug: SCY-078 plus DAB

INTERVENTIONS:
Drug: DAB — Single oral 150-mg dose of DAB on Day 1 AM.
  Arms: Treatment A
Drug: SCY-078 plus DAB — Twice daily (BID), every 12 hours (Q12H) oral doses of SCY-078 750 mg on Day 1 and Day 2; and single oral AM doses of SCY-078 750 mg on Day 3 and Day 4. On Day 3 a single 150-mg dose of DAB will be administered one hour after the AM dose of SCY-078.
  Arms: Treatment B

SUMMARY:
This is a Phase 1 open-label, randomized, two-period, crossover study to evaluate the effect of repeated oral doses of SCY-078 (Ibrexafungerp) on the pharmacokinetics of dabigatran administered orally to healthy subjects.

DETAILED DESCRIPTION:
The two-period crossover study will consist of two treatments administered in random order. Treatments will be separated by a minimum of 10 day wash-out (between last dose in the first period and first dose in the subsequent period). Healthy male and female subjects will will be enrolled to assess the effects on a single dose of dabigatran mesylate (DAB).

Subjects will be screened within 4 weeks prior to dosing and randomized to a treatment sequence (AB or BA) in a crossover fashion.

Treatment A: Single oral 150mg dose of DAB. Treatment B: Twice daily (BID), every 12 hours (Q12H) oral doses of SCY-078 750mg on Day and Day 2; and single oral AM doses of SCY-078 750mg on Day 3 and Day. On Day 3, a single 150mg dose of DAB will be administered 1 hour after the AM dose of SCY-078.

Subjects will fast overnight after being admitted to the clinic on Day -1 and will remain in the clinic until the final procedures are complete.

Twenty eight male and female subjects between 18 and 55 years (inclusive) will be enrolled into the study. Subjects who discontinue may be replaced.

ELIGIBILITY:
Inclusion Criteria:

1. is a male or female between 18 to 55 years, inclusive, of age at the prestudy (screening) visit (time of signing the Informed Consent).
2. has a Body Mass Index (BMI) 18.0 - 32 kg/m2 at the prestudy (screening) visit. BMI is calculated by taking the subject's weight in kg and dividing by the subject's height in meters, squared.
3. is judged to be in good physical and mental health based on medical history, physical examination, vital sign measurements, ECG, and laboratory safety tests performed at the prestudy (screening) visit and/or prior to administration of the initial dose of study drug. Subjects will be enrolled at the discretion of the investigator.
4. is a nonsmoker and has not used nicotine or nicotine containing products for 6 months prior to screening.
5. is willing and able to sign the informed consent and understands the study procedures and agrees to comply with all restrictions and participate in the study.
6. is not pregnant or lactating (for women of childbearing potential) and must agree to use adequate double barrier birth control.

Exclusion Criteria:

1. has a contra-indication to PRADAXA® (dabigatran etexilate mesylate)
2. has a prior history of convulsions, or hemorrhagic disease
3. has a history of peptic ulcer disease that is currently being treated.
4. is pregnant or is lactating
5. has a history of uncontrolled or unstable cardiovascular, respiratory, renal, hepatic, gastrointestinal, endocrine, hematopoietic, neoplastic, and/or neurological disease.
6. has had any major surgery within 30 days of dosing with study drug.
7. has consumed Seville or blood oranges, grapefruit or grapefruit juice, or mulberry juice as well as vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, and mustard) or charbroiled meats from 4 days prior to the dose of study medication.
8. has consumed any alcohol within 7 days prior to the dose of study medication.
9. is a smoker or has used tobacco or any nicotine-containing products within the 6 months prior to screening.
10. has a positive test result for drugs of abuse, alcohol, or cotinine at screening or before dosing.
11. has participated in a clinical investigation of any drug, biological, or other investigational therapy, device or procedure 30 days before dosing
12. has a history of an allergic reaction to SCY-078 or any of its excipients. or is allergic to PRADAXA® (dabigatran etexilate mesylate), or its inactive ingredients.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of DAB administered with SCY-078, AUC | 17 days
  AUC0-48 of DAB when taken with SCY-078

SECONDARY OUTCOMES:
Pharmacokinetics of DAB administered with SCY-078, Cmax | 17 days
  Cmax DAB when taken with SCY-078.
Pharmacokinetics of DAB administered with SCY-078, Tmax | 17 days
  Tmax of DAB when taken with SCY-078.
Pharmacokinetics of DAB administered with SCY-078, Half Life | 17 Days
  Half Life of DAB when taken with SCY-078.
Safety and tolerability of oral dosing of combination of DAB with SCY-078 | 7 weeks
  Incidence of treatment-related adverse events (AE) and discontinuations due to (AEs)

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX, Adelaide, South Australia, Australia